CLINICAL TRIAL: NCT03122223
Title: A Phase 1/2a Clinical Trial to Evaluate the Safety and Immunogenicity of ALVAC-HIV (vCP2438) and of MF59®- or AS01B-adjuvanted Clade C Env Protein, in Healthy, HIV-uninfected Adult Participants
Brief Title: Evaluating the Safety and Immunogenicity of ALVAC-HIV and MF59®- or AS01B-adjuvanted Bivalent Subtype C gp120 in Healthy, HIV-uninfected Adult Participants
Acronym: HVTN 120
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: GlaxoSmithKline (Industry); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 120; 36128 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-02-14; First posted 2017-04-20 (Actual); Results first posted 2021-01-08 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- ALVAC-HIV + 100mcg Protein/MF59 + Placebo (Active Comparator): 50 participants will receive 1 mL ALVAC-HIV injection in the left deltoid on Months 0, 1, 3, and 6. They will receive 0.5 mL100 mcg Protein/MF59 and 0.75 mL placebo injection in the right deltoid on Months 3 and 6.
  Interventions: Biological: ALVAC-HIV (vCP2438); Biological: Bivalent subtype C gp120/MF59; Biological: Placebo
- ALVAC-HIV + 100mcg Protein/AS01(B) + Placebo (Active Comparator): 50 participants will receive 1 mL ALVAC-HIV injection in the left deltoid on Months 0, 1, 3, and 6. They will receive 0.75 mL100 mcg Protein/AS01(B) and 0.5 mL placebo injection in the right deltoid on Months 3 and 6.
  Interventions: Biological: ALVAC-HIV (vCP2438); Biological: Bivalent subtype C gp120/AS01(B); Biological: Placebo
- ALVAC-HIV + 20mcg Protein/AS01(B) + Placebo (Active Comparator): 50 participants will receive 1 mL ALVAC-HIV injection in the left deltoid on Months 0, 1, 3, and 6. They will receive 0.75 mL 20 mcg Protein/AS01(B) and 0.5 mL placebo injection in the right deltoid on Months 3 and 6.
  Interventions: Biological: ALVAC-HIV (vCP2438); Biological: Bivalent subtype C gp120/AS01(B); Biological: Placebo
- Placebo (Placebo Comparator): 10 participants will receive 1 mL of the placebo injection in the left deltoid on Months 0, 1, 3, and 6. They will receive 0.5 mL of the placebo injection and 0.75 mL of a separate placebo injection in the right deltoid on Months 3 and 6.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ALVAC-HIV (vCP2438) — expresses the gene products 96ZM651 gp120 (clade C strain) linked to the sequences encoding the HIV-1 transmembrane anchor (TM) sequence of gp41 (28 amino acids clade B LAI strain) and Gag and Pro (clade B LAI strain). It is formulated as a lyophilized vaccine for injection at a viral titer greater than or equal to 1 × 10^6 cell culture infectious dose (CCID)50 and less than 1 × 10^8 CCID50 (nominal dose of 10^7 CCID50) and is reconstituted with 1 mL of sterile sodium chloride solution (NaCl 0.4%), administered IM as a single 1 mL dose.
  Arms: ALVAC-HIV + 100mcg Protein/AS01(B) + Placebo; ALVAC-HIV + 100mcg Protein/MF59 + Placebo; ALVAC-HIV + 20mcg Protein/AS01(B) + Placebo
Biological: Bivalent subtype C gp120/MF59 — clade C TV1.C gp120 Env and clade C 1086.C gp120 Env, each at a dose of 100 mcg, mixed with MF59 adjuvant, administered IM as a single 0.5 mL dose.
  Arms: ALVAC-HIV + 100mcg Protein/MF59 + Placebo
Biological: Bivalent subtype C gp120/AS01(B) — clade C TV1.C gp120 Env and clade C 1086.C gp120 Env, each at a dose of 20 mcg or 100 mcg, mixed with AS01B adjuvant, administered IM as a single 0.75 mL dose.
  Arms: ALVAC-HIV + 100mcg Protein/AS01(B) + Placebo; ALVAC-HIV + 20mcg Protein/AS01(B) + Placebo
Biological: Placebo — Sodium Chloride for Injection, 0.9%, administered IM.

SUMMARY:
A phase 1/2a clinical trial to evaluate the safety and immunogenicity of ALVAC-HIV (vCP2438) and of MF59®- or AS01B-adjuvanted clade C Env protein, in healthy, HIV-uninfected adult participants

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of ALVAC-HIV and bivalent gp120 protein/MF59 or bivalent gp120 protein/AS01(B). This study will also compare HIV-specific CD4+ T-cell response rates at the Month 6.5 timepoint (2 weeks after the fourth vaccination) of ALVAC-HIV and bivalent gp120 protein/MF59 to each of the bivalent gp120 protein/AS01(B) vaccine regimens. Additionally, this study will compare HIV-specific Env-gp120 binding antibody response magnitudes at the Month 12 timepoint (6 months after the fourth vaccination) of ALVAC-HIV and bivalent gp120 protein/MF59 to each of the bivalent gp120 protein/AS01(B) vaccine regimens.

The study will enroll 160 healthy, HIV-uninfected volunteers aged 18 to 40 years. Groups 1 to 3 will consist of a total of 150 participants who will receive the vaccines at Months 0, 1, 3, and 6, while 10 participants in Group 4 will receive placebos at Months 0, 1, 3, 6.

Study visits will include a physical examination, an interview and/or questionnaire, HIV testing and HIV risk-reduction counseling, and urine and blood collection. Participants may optionally choose to provide rectal fluid, cervical fluid, semen, and/or stool samples.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria:

* Age of 18 to 40 years
* Access to a participating HVTN clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; provides answers to a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent before the last required clinic visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit (see the study protocol for more information about low risk guidelines).

Laboratory Inclusion Values:

Hemogram/Complete Blood Count (CBC):

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were assigned female sex at birth, greater than or equal to 13.0 g/dL for volunteers who were assigned male sex at birth. For transgender participants who have been on hormone therapy for more than 6 consecutive months, determine hemoglobin eligibility based on the gender with which they identify (ie, a transgender female who has been on hormone therapy for more than 6 consecutive months should be assessed for eligibility using the hemoglobin parameters for persons assigned female sex at birth).
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry:

* Chemistry panel: ALT, AST, and ALP less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal.

Virology:

* Negative HIV-1 and -2 blood test: US volunteers must have a negative FDA-approved enzyme immunoassay (EIA). Non-US sites may use locally available assays that have been approved by HVTN Laboratory Operations.
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine:

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

Reproductive Status:

* Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: Africa - A volunteer who was assigned female sex at birth must:

  * Agree to consistently use effective contraception (see the study protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception for participants in Africa is defined as using 2 methods of birth control. These include 1 of the following methods:

    * Condoms (male or female), or
    * Diaphragm or cervical cap, PLUS 1 of the following methods:
    * Intrauterine device (IUD),
    * Hormonal contraception (in accordance with applicable national contraception guidelines),
    * Successful vasectomy in any partner assigned male at birth (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity after vasectomy); or
    * Any other contraceptive method approved by the HVTN 120 Protocol Safety Review Team (PSRT)
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Reproductive status: United States - A volunteer who was assigned female sex at birth must:

  * Agree to consistently use effective contraception (see the study protocol for more information) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception for participants in the United States is defined as using any 1 or more of the following methods of birth control:

    * Condoms (male or female) with or without spermicide,
    * Diaphragm or cervical cap with spermicide,
    * Intrauterine device (IUD),
    * Hormonal contraception, or
    * Successful vasectomy in any partner assigned male at birth (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity after vasectomy); or
    * Any other contraceptive method approved by the HVTN 120 PSRT
  * Or must not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or must be sexually abstinent.
* Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Other:

* Volunteers 21 years of age and older who were assigned female sex at birth consenting to provide cervical samples:

  * Pap smear within:

    * the 3 years prior to enrollment with the latest result reported as normal or ASCUS (atypical squamous cells of undetermined significance), OR
    * the 5 years prior to enrollment, with the latest result reported as normal, or ASCUS with no evidence of high risk HPV.
  * If no pap smear was done within the last 3 years prior to enrollment (or within the last 5 years, if high risk HPV testing was performed), the volunteer must be willing to undergo a pap smear with the result reported as normal or ASCUS prior to sample collection.

Exclusion Criteria:

General:

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 120 study
* Pregnant or breastfeeding
* Active duty and reserve U.S. military personnel

Vaccines and Other Injections:

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 120 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of monoclonal antibodies (mAbs), whether licensed or investigational; the HVTN 120 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 120 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) more than 5 years ago, eligibility for enrollment will be determined by the HVTN 120 PSRT on a case-by-case basis.
* Live attenuated vaccines received within 30 days before first study vaccination or scheduled within 14 days after first study vaccination (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever; live attenuated influenza vaccine)
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first study vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first study vaccination or that are scheduled within 14 days after first study vaccination

Immune System:

* Immunosuppressive medications received within 168 days before first study vaccination. (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral prednisone or equivalent at doses less than or equal to 60 mg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment.
* Serious adverse reactions to vaccines or to vaccine components such as eggs, egg products, or neomycin, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first study vaccination (for mAb see criterion above)
* Autoimmune disease
* Immunodeficiency

Clinically Significant Medical Conditions:

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent US National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
* In the past year has either of the following:

  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2. (Not excluded: type 2 cases controlled with diet alone or a history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Z Mike Chirenje, Study Chair — UZ-UCSF Collaborative Research Program
Locations (12):
- United States (9):
  - Bridge HIV CRS, San Francisco, California
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Case Clinical Research Site, Cleveland, Ohio
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington
- National Institute for Medical Research (NIMR) - Mbeya Medical Research Center (MMRC) Network CRS, Mbeya, Tanzania
- Matero Reference Clinic CRS, Lusaka, Zambia
- Seke South CRS, Chitungwiza, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Chirenje ZM, Laher F, Dintwe O, Muyoyeta M, deCamp AC, He Z, Grunenberg N, Laher Omar F, Seaton KE, Polakowski L, Woodward Davis AS, Maganga L, Baden LR, Mayer K, Kalams S, Keefer M, Edupuganti S, Rodriguez B, Frank I, Scott H, Stranix-Chibanda L, Gurunathan S, Koutsoukos M, Van Der Meeren O, DiazGranados CA, Paez C, Andersen-Nissen E, Kublin J, Corey L, Ferrari G, Tomaras G, McElrath MJ. Protein Dose-Sparing Effect of AS01B Adjuvant in a Randomized Preventive HIV Vaccine Trial of ALVAC-HIV (vCP2438) and Adjuvanted Bivalent Subtype C gp120. J Infect Dis. 2024 Aug 16;230(2):e405-e415. doi: 10.1093/infdis/jiad434. PMID 37795976

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine w/ MF59: ALVAC-HIV at Months 0 and 1, ALVAC-HIV + 100mcg Protein/MF59 at Months 3 and 6
- Vaccine w/ AS01B - High Dose: ALVAC-HIV at Months 0 and 1, ALVAC-HIV + 100mcg Protein/AS01B at Months 3 and 6
- Vaccine w/ AS01B - Low Dose: ALVAC-HIV at Months 0 and 1, ALVAC-HIV + 20mcg Protein/AS01B at Months 3 and 6
- Placebo: Placebo at Months 0, 1, 3, and 6
Period: Overall Study
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Started | 50 | 50 | 50 | 10
Month 6.5 Immunogenicity Cohort | 49 | 48 | 47 | 8
Month 12 Immunogenicity Cohort | 47 | 45 | 46 | 10
Completed | 47 | 45 | 46 | 10
Not Completed | 3 | 5 | 4 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 2 | 0
Not completed — Participant unable to adhere | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 50 | 10 | 160
Age, Continuous [Median (Full Range); unit: years] | 24 [19 to 40] | 23.5 [18 to 38] | 25.5 [19 to 39] | 24 [18 to 37] | 24 [18 to 40]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0
  18 - 20 years | 9 | 9 | 6 | 2 | 26
  21 - 30 years | 30 | 32 | 32 | 6 | 100
  31 - 40 years | 11 | 9 | 12 | 2 | 34
  41 - 50 years | 0 | 0 | 0 | 0 | 0
  Above 50 years | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 25 | 2 | 88
  Male | 19 | 20 | 25 | 8 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 1 | 5
  Not Hispanic or Latino | 48 | 49 | 49 | 9 | 155
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 30 | 31 | 31 | 7 | 99
  White | 17 | 16 | 17 | 3 | 53
  More than one race | 2 | 3 | 1 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 20 | 20 | 20 | 4 | 64
  Tanzania | 15 | 15 | 15 | 3 | 48
  Zambia | 5 | 5 | 5 | 1 | 16
  Zimbabwe | 10 | 10 | 10 | 2 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms During the Vaccine Regimen
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017. The maximum grade observed for each symptom over the time frame is presented;
Time Frame: Measured through 7 days after participants' last vaccination at Month 0,1,3, and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 10
Participants
  Pain: None | 16 | 18 | 16 | 7
  Pain: Mild | 27 | 17 | 20 | 3
  Pain: Moderate | 6 | 13 | 14 | 0
  Pain: Severe | 1 | 2 | 0 | 0
  Pain: Potentially Life-threatening | 0 | 0 | 0 | 0
  Tenderness: None | 21 | 20 | 15 | 8
  Tenderness: Mild | 22 | 12 | 18 | 2
  Tenderness: Moderate | 6 | 17 | 17 | 0
  Tenderness: Severe | 1 | 1 | 0 | 0
  Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Pain and/or Tenderness: None | 15 | 15 | 12 | 7
  Pain and/or Tenderness: Mild | 26 | 17 | 19 | 3
  Pain and/or Tenderness: Moderate | 8 | 16 | 19 | 0
  Pain and/or Tenderness: Severe | 1 | 2 | 0 | 0
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0 | 0 | 0
  Erythema: None | 46 | 42 | 43 | 9
  Erythema: Mild | 2 | 2 | 0 | 1
  Erythema: Moderate | 2 | 2 | 6 | 0
  Erythema: Severe | 0 | 4 | 1 | 0
  Erythema: Potentially Life-threatening | 0 | 0 | 0 | 0
  Induration: None | 49 | 45 | 43 | 10
  Induration: Mild | 0 | 1 | 3 | 0
  Induration: Moderate | 1 | 1 | 4 | 0
  Induration: Severe | 0 | 3 | 0 | 0
  Induration: Potentially Life-threatening | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 45 | 42 | 39 | 9
  Erythema and/or Induration: Mild | 2 | 2 | 2 | 1
  Erythema and/or Induration: Moderate | 3 | 2 | 8 | 0
  Erythema and/or Induration: Severe | 0 | 4 | 1 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms During the Primary Vaccine Regimen
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1,July 2017. The maximum grade observed for each symptom over the time frame is presented;
Time Frame: Measured through 7 days after each vaccination at Month 0, 1, 3, and 6
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 10
Participants
  Malaise and/or fatigue: None | 26 | 27 | 22 | 6
  Malaise and/or fatigue: Mild | 17 | 7 | 12 | 3
  Malaise and/or fatigue: Moderate | 6 | 13 | 12 | 1
  Malaise and/or fatigue: Severe | 1 | 3 | 4 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0
  Myalgia: None | 38 | 32 | 29 | 7
  Myalgia: Mild | 11 | 7 | 9 | 2
  Myalgia: Moderate | 1 | 9 | 8 | 1
  Myalgia: Severe | 0 | 2 | 4 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Headache: None | 30 | 26 | 25 | 7
  Headache: Mild | 15 | 13 | 15 | 1
  Headache: Moderate | 5 | 11 | 7 | 2
  Headache: Severe | 0 | 0 | 3 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0
  Nausea: None | 42 | 39 | 38 | 7
  Nausea: Mild | 6 | 10 | 7 | 3
  Nausea: Moderate | 2 | 1 | 5 | 0
  Nausea: Severe | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0
  Vomiting: None | 48 | 48 | 49 | 9
  Vomiting: Mild | 1 | 2 | 0 | 1
  Vomiting: Moderate | 1 | 0 | 1 | 0
  Vomiting: Severe | 0 | 0 | 0 | 0
  Vomiting: Potentially Life-threatening | 0 | 0 | 0 | 0
  Chills: None | 42 | 33 | 30 | 10
  Chills: Mild | 7 | 10 | 8 | 0
  Chills: Moderate | 1 | 6 | 10 | 0
  Chills: Severe | 0 | 1 | 2 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0
  Arthralgia: None | 40 | 39 | 35 | 7
  Arthralgia: Mild | 7 | 3 | 5 | 3
  Arthralgia: Moderate | 3 | 7 | 10 | 0
  Arthralgia: Severe | 0 | 1 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 20 | 21 | 18 | 4
  Max. Systemic Symptoms: Mild | 18 | 10 | 13 | 4
  Max. Systemic Symptoms: Moderate | 11 | 16 | 14 | 2
  Max. Systemic Symptoms: Severe | 1 | 3 | 5 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0
  Temperature: None | 47 | 46 | 45 | 10
  Temperature: Mild | 2 | 2 | 5 | 0
  Temperature: Moderate | 1 | 2 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0

3. Primary Outcome: Frequency of Adverse Events by Relationship to the Study Product
Description: For participants reporting multiple AEs over the time frame, the maximum relationship is counted.
Time Frame: Measured through 30 days after each vaccination at Month 0, 1, 3 and 6.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 10
Participants
  Related | 2 | 7 | 2 | 0
  Not Related | 30 | 21 | 24 | 6
  No AE Reported | 18 | 22 | 24 | 4

4. Primary Outcome: Frequency of SAEs, AESIs, and New Chronic Conditions
Description: No SAEs, AESIs, or new chronic conditions were reported over the course of the study
Time Frame: Measured through Month 18.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 10
Participants
  SAE | 0 | 0 | 0 | 0
  AESI or new Chronic Condiiton | 0 | 0 | 0 | 0
  No SAE or AESI or New Chronic condition | 50 | 50 | 50 | 10

5. Primary Outcome: Alkaline Phosphatase, AST, ALT in U/L
Description: Laboratory results are summarized by analyte and timepoint.
Time Frame: Measured at Month 0 (Screening) ,0.5(Day 14), 1.5 (Day 42) , 3.5 (Day 98) and 6.5 (Day 182)
Population: The "overall number of participants analyzed" represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, or they missed the scheduled visit, or they terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 10
U/L
  Alkaline Phosphatase (U/L)- Screening | 75 [60 to 101] | 69 [55 to 94] | 72 [63 to 92] | 78 [63 to 103]
  Alkaline Phosphatase (U/L)- Day14: number analyzed (Participants) | 50 | 49 | 48 | 10
  Alkaline Phosphatase (U/L)- Day14 | 74.5 [55 to 94] | 67 [55 to 85] | 70 [56.5 to 87.5] | 78 [55 to 88]
  Alkaline Phosphatase (U/L)- Day42: number analyzed (Participants) | 48 | 49 | 49 | 9
  Alkaline Phosphatase (U/L)- Day42 | 70 [57.5 to 93] | 65 [52 to 87] | 67 [60 to 88] | 77 [61 to 88]
  Alkaline Phosphatase (U/L)- Day98: number analyzed (Participants) | 48 | 48 | 50 | 8
  Alkaline Phosphatase (U/L)- Day98 | 70.5 [58 to 90] | 67 [51 to 90] | 69.5 [60 to 84] | 81.5 [60.5 to 93.5]
  Alkaline Phosphatase (U/L)- Day182: number analyzed (Participants) | 49 | 48 | 47 | 8
  Alkaline Phosphatase (U/L)- Day182 | 72 [58 to 88] | 66.5 [50 to 82.5] | 68 [55 to 82] | 74.5 [54 to 90]
  AST (U/L)- Screening | 20.5 [16 to 24] | 20 [16 to 24] | 22 [17 to 26] | 22.5 [18 to 26]
  AST (U/L)- Day14: number analyzed (Participants) | 50 | 49 | 48 | 10
  AST (U/L)- Day14 | 20 [16 to 24] | 20 [17 to 23] | 21 [17 to 24] | 21.5 [19 to 24]
  AST (U/L)- Day42: number analyzed (Participants) | 48 | 49 | 50 | 9
  AST (U/L)- Day42 | 22 [16 to 25.5] | 21 [18 to 24] | 20 [16 to 26] | 21 [19 to 22]
  AST (U/L)- Day98: number analyzed (Participants) | 48 | 48 | 50 | 8
  AST (U/L)- Day98 | 21 [16 to 25.5] | 20 [17.5 to 23] | 20 [18 to 24] | 25.5 [18 to 28]
  AST (U/L)- Day182: number analyzed (Participants) | 49 | 48 | 47 | 8
  AST (U/L)- Day182 | 22 [17 to 26] | 19 [17 to 23.5] | 20 [16 to 25] | 25.5 [18.5 to 30.5]
  ALT (SGPT) (U/L)- Screening | 17.5 [14 to 22] | 16.5 [13 to 24] | 16.5 [12 to 22] | 18.5 [16 to 26]
  ALT (SGPT) (U/L)- Day14: number analyzed (Participants) | 50 | 49 | 48 | 10
  ALT (SGPT) (U/L)- Day14 | 17 [13 to 21] | 16 [13 to 21] | 16.5 [12 to 21] | 20.5 [17 to 22]
  ALT (SGPT) (U/L)- Day42: number analyzed (Participants) | 48 | 49 | 50 | 9
  ALT (SGPT) (U/L)- Day42 | 17 [13 to 22] | 18 [13 to 25] | 16 [12 to 23] | 19 [17 to 21]
  ALT (SGPT) (U/L)- Day98: number analyzed (Participants) | 48 | 48 | 50 | 8
  ALT (SGPT) (U/L)- Day98 | 16.5 [12 to 22] | 18 [13 to 23] | 16.5 [12 to 21] | 24 [15 to 32]
  ALT (SGPT) (U/L)- Day182: number analyzed (Participants) | 49 | 48 | 47 | 8
  ALT (SGPT) (U/L)- Day182 | 16 [13 to 21] | 17.5 [12 to 24] | 17 [13 to 21] | 22.5 [17 to 28.5]

6. Primary Outcome: Hemoglobin, Creatinine in g/dL
Description: Laboratory results are summarized by analyte and timepoint.
Time Frame: Measured at Month 0 (Screening) ,0.5(Day 14), 1.5 (Day 42) , 3.5 (Day 98) and 6.5 (Day 182)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 10
g/dL
  Hemoglobin (g/dL)- Screening | 14.45 [13.4 to 15.7] | 15.05 [13.6 to 16.4] | 14.7 [13.4 to 16.4] | 14.9 [14.7 to 16.1]
  Hemoglobin (g/dL)- Day14: number analyzed (Participants) | 50 | 49 | 48 | 10
  Hemoglobin (g/dL)- Day14 | 14.1 [12.9 to 15.7] | 14.5 [13.2 to 16.1] | 14 [12.95 to 15.5] | 14.9 [14.1 to 15.2]
  Hemoglobin (g/dL)- Day42: number analyzed (Participants) | 48 | 49 | 50 | 9
  Hemoglobin (g/dL)- Day42 | 14.45 [13.2 to 15.25] | 14.6 [13.5 to 16.1] | 14.05 [12.9 to 16] | 14.8 [14.6 to 15]
  Hemoglobin (g/dL)- Day98: number analyzed (Participants) | 48 | 48 | 50 | 8
  Hemoglobin (g/dL)- Day98 | 14.5 [13.2 to 15.55] | 14.8 [13.8 to 16.25] | 14.1 [13.3 to 16.3] | 14.45 [14.1 to 15.45]
  Hemoglobin (g/dL)- Day182: number analyzed (Participants) | 49 | 48 | 47 | 8
  Hemoglobin (g/dL)- Day182 | 14 [12.8 to 14.8] | 14.25 [13.3 to 15.95] | 14 [12.7 to 15.5] | 14.45 [14 to 15.95]
  Creatinine (g/dL)- Screening | 0.00073 [0.00061 to 0.00087] | 0.00079 [0.00068 to 0.0009] | 0.000785 [0.00069 to 0.00089] | 0.00086 [0.00074 to 0.00097]
  Creatinine (g/dL)- Day14: number analyzed (Participants) | 50 | 49 | 49 | 10
  Creatinine (g/dL)- Day14 | 0.00076 [0.00066 to 0.00085] | 0.0008 [0.00068 to 0.00086] | 0.00076 [0.0007 to 0.00086] | 0.000765 [0.0007 to 0.00091]
  Creatinine (g/dL)- Day42: number analyzed (Participants) | 48 | 49 | 50 | 9
  Creatinine (g/dL)- Day42 | 0.00075 [0.000615 to 0.00086] | 0.00075 [0.00064 to 0.00086] | 0.0008 [0.0007 to 0.00087] | 0.00081 [0.0007 to 0.00084]
  Creatinine (g/dL)- Day98: number analyzed (Participants) | 48 | 48 | 50 | 8
  Creatinine (g/dL)- Day98 | 0.000775 [0.000665 to 0.00086] | 0.000775 [0.000685 to 0.000835] | 0.0008 [0.0007 to 0.0009] | 0.000885 [0.000765 to 0.00095]
  Creatinine (g/dL)- Day182: number analyzed (Participants) | 49 | 48 | 47 | 8
  Creatinine (g/dL)- Day182 | 0.00071 [0.00066 to 0.0009] | 0.0008 [0.0007 to 0.00086] | 0.0008 [0.0007 to 0.00088] | 0.000895 [0.0007 to 0.00102]

7. Primary Outcome: WBC, Platelets, Lymphocytes, Neutrophils in Thousand Cells/Cubic mm
Description: Laboratory results are summarized by analyte and timepoint.
Time Frame: Measured at Month 0 (Screening) ,0.5(Day 14), 1.5 (Day 42) , 3.5 (Day 98) and 6.5 (Day 182)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: thousand cells/cubic mm
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 10
thousand cells/cubic mm
  WBC (1000/cubic mm)- Screening | 5.29 [4.43 to 6.54] | 5.92 [5 to 6.8] | 5.4 [4.53 to 6.5] | 5.125 [4.11 to 5.9]
  WBC (1000/cubic mm)- Day14: number analyzed (Participants) | 50 | 49 | 48 | 10
  WBC (1000/cubic mm)- Day14 | 5.3 [4.1 to 6.7] | 5.8 [4.3 to 6.81] | 5.535 [4.22 to 6.4] | 4.94 [4.36 to 5.2]
  WBC (1000/cubic mm)- Day42: number analyzed (Participants) | 48 | 49 | 50 | 9
  WBC (1000/cubic mm)- Day42 | 5.065 [4.375 to 6.405] | 5.28 [4.4 to 6.5] | 5.025 [3.9 to 6.2] | 4.58 [4.1 to 5.3]
  WBC (1000/cubic mm)- Day98: number analyzed (Participants) | 48 | 48 | 50 | 8
  WBC (1000/cubic mm)- Day98 | 4.805 [4.355 to 5.645] | 5.33 [4.35 to 6.85] | 5.15 [4.36 to 6.6] | 4.79 [3.475 to 7.085]
  WBC (1000/cubic mm)- Day182: number analyzed (Participants) | 49 | 48 | 47 | 8
  WBC (1000/cubic mm)- Day182 | 4.93 [4.23 to 6.59] | 5.36 [4.305 to 6.67] | 5.28 [4.01 to 6.98] | 5.28 [4.74 to 5.68]
  Platelets (1000/cubic mm)- Screening | 263.5 [220 to 297] | 263.5 [209 to 301] | 233 [215 to 275] | 223.5 [211 to 280]
  Platelets (1000/cubic mm)- Day14: number analyzed (Participants) | 50 | 49 | 48 | 10
  Platelets (1000/cubic mm)- Day14 | 264 [226 to 303] | 248 [222 to 297] | 238 [214 to 279] | 236.5 [222 to 247]
  Platelets (1000/cubic mm)- Day42: number analyzed (Participants) | 48 | 49 | 50 | 9
  Platelets (1000/cubic mm)- Day42 | 254 [224.5 to 283.5] | 266 [213 to 316] | 242.5 [207 to 270] | 234 [230 to 265]
  Platelets (1000/cubic mm)- Day98: number analyzed (Participants) | 48 | 48 | 50 | 8
  Platelets (1000/cubic mm)- Day98 | 264.5 [223.5 to 293] | 267 [214.5 to 304] | 246.5 [202 to 292] | 221 [187.5 to 275.5]
  Platelets (1000/cubic mm)- Day182: number analyzed (Participants) | 49 | 48 | 47 | 8
  Platelets (1000/cubic mm)- Day182 | 264 [239 to 293] | 260 [224.5 to 308.5] | 251.1 [218 to 301] | 245.5 [193 to 315]
  Lymphocytes (1000/cubic mm)- Screening | 1.935 [1.59 to 2.31] | 2.014 [1.67 to 2.361] | 1.84 [1.56 to 2.4] | 1.9455 [1.58 to 2.32]
  Lymphocytes (1000/cubic mm)- Day14: number analyzed (Participants) | 50 | 49 | 48 | 10
  Lymphocytes (1000/cubic mm)- Day14 | 1.825 [1.578 to 2.29] | 1.98 [1.647 to 2.593] | 1.7945 [1.5855 to 2.231] | 1.705 [1.2 to 2.01]
  Lymphocytes (1000/cubic mm)- Day42: number analyzed (Participants) | 48 | 49 | 50 | 9
  Lymphocytes (1000/cubic mm)- Day42 | 1.9135 [1.5945 to 2.319] | 1.88 [1.62 to 2.25] | 1.7995 [1.498 to 2.12] | 1.668 [1.36 to 1.97]
  Lymphocytes (1000/cubic mm)- Day98: number analyzed (Participants) | 48 | 48 | 50 | 8
  Lymphocytes (1000/cubic mm)- Day98 | 1.86 [1.5805 to 2.314] | 1.99 [1.625 to 2.231] | 1.812 [1.532 to 2.18] | 1.7145 [1.346 to 2.475]
  Lymphocytes (1000/cubic mm)- Day182: number analyzed (Participants) | 49 | 48 | 47 | 8
  Lymphocytes (1000/cubic mm)- Day182 | 1.913 [1.65 to 2.27] | 1.91 [1.556 to 2.2505] | 1.767 [1.447 to 2.265] | 1.7905 [1.54 to 2.585]
  Neutrophils (1000/cubic mm)- Screening | 2.6835 [2.13 to 3.64] | 2.9995 [2.499 to 4.18] | 2.8925 [2.211 to 3.87] | 2.415 [2.207 to 3.02]
  Neutrophils (1000/cubic mm)- Day14: number analyzed (Participants) | 50 | 49 | 48 | 10
  Neutrophils (1000/cubic mm)- Day14 | 2.8755 [1.936 to 3.866] | 3.07 [2.08 to 3.79] | 2.896 [2.0355 to 3.5425] | 2.529 [2.44 to 3.38]
  Neutrophils (1000/cubic mm)- Day42: number analyzed (Participants) | 48 | 49 | 50 | 9
  Neutrophils (1000/cubic mm)- Day42 | 2.577 [2.02 to 3.75] | 2.82 [2.023 to 3.47] | 2.662 [1.914 to 3.441] | 2.55 [2.013 to 2.86]
  Neutrophils (1000/cubic mm)- Day98: number analyzed (Participants) | 48 | 48 | 50 | 8
  Neutrophils (1000/cubic mm)- Day98 | 2.37 [2.053 to 2.954] | 2.605 [1.818 to 3.988] | 2.66 [2.176 to 3.709] | 2.105 [1.6215 to 4.06]
  Neutrophils (1000/cubic mm)- Day182: number analyzed (Participants) | 49 | 48 | 47 | 8
  Neutrophils (1000/cubic mm)- Day182 | 2.66 [1.884 to 3.29] | 2.776 [2.23 to 3.7575] | 2.98 [2.01 to 4] | 2.45 [2.355 to 3.22]

8. Primary Outcome: AEs or Reactro Leading to Early Participant Withdrawal or Early Discontinuation of Study Products Administration Throughout the Study.
Description: From the study product discontinuation form, study product administration reasons are tabulated by treatment arm
Time Frame: Measured through month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 10
Participants
  Clinical Event | 0 | 0 | 0 | 0
  Reactogenicity | 0 | 0 | 1 | 0
  Other reason | 1 | 2 | 1 | 0
  No discontinuation | 49 | 48 | 48 | 10

9. Primary Outcome: Occurrence of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine, After the Primary Vaccine Regimen. Measured by Flow Cytometry.
Description: PBMC samples are stimulated with synthetic peptide pools or left unstimulated as a negative control. For each sample, T-cell subset, and peptide pool, response magnitude is % cells expressing IL-2/IFNy after peptide stimulation minus % cells expressing markers after no stimulation. A contingency table is constructed to assess response: stimulation (peptide/none) vs. marker expression (yes/no). A one-sided Fisher's exact test is applied, testing if the number of cells positive for the marker is equal in the stimulated vs. unstimulated cells. A discrete Bonferroni adjustment is made over the peptide pools. A response is positive if p<=0.00001.The number and percentage of participants with positive responses are summarized by peptide pool.
Time Frame: Measured at Month 6.5
Population: In this report, the "overall number of participants analyzed" represents the HIV uninfected participants with specimens at Month6.5. The "Number Analyzed" in the Outcome Measure Data Table shows the number of participants with available ICS data after filtering for assay specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 49 | 48 | 47 | 8
Participants
  1086 gp120: number analyzed (Participants) | 42 | 42 | 38 | 7
  1086 gp120 | 18 | 38 | 35 | 0
  Env-1-ZM96: number analyzed (Participants) | 42 | 41 | 38 | 7
  Env-1-ZM96 | 19 | 34 | 37 | 0
  Env-2-ZM96: number analyzed (Participants) | 42 | 42 | 38 | 7
  Env-2-ZM96 | 6 | 17 | 16 | 0
  LAI Gag: number analyzed (Participants) | 42 | 42 | 38 | 7
  LAI Gag | 0 | 4 | 1 | 0
  LAI gp41TM: number analyzed (Participants) | 42 | 42 | 38 | 7
  LAI gp41TM | 1 | 0 | 1 | 0
  TV1 gp120: number analyzed (Participants) | 42 | 42 | 38 | 7
  TV1 gp120 | 23 | 39 | 37 | 0

10. Primary Outcome: Level of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine, After the Primary Vaccine Regimen. Measured by Flow Cytometry.
Description: Measured by flow cytometry ICS assay: refer to earlier description for assay methods and analysis variable derivation. The percentage of T-cells expressing IL-1/IFNy are summarized for positive responders only.
Time Frame: Measured at Month 6.5
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: % CD4+ T-cells
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 49 | 48 | 47 | 8
% CD4+ T-cells
  1086 gp120: number analyzed (Participants) | 42 | 42 | 38 | 7
  1086 gp120 | 0.043625715 [0.01686033 to 0.14821546] | 0.21257737 [0.13504277 to 0.3292746] | 0.236469065 [0.18752656 to 0.50737339] | -0.00430092 [-0.00747952 to 0.0069845]
  Env-1-ZM96: number analyzed (Participants) | 42 | 41 | 38 | 7
  Env-1-ZM96 | 0.045957505 [0.01215409 to 0.11491243] | 0.17245457 [0.08842416 to 0.26856661] | 0.204674615 [0.12129456 to 0.33604536] | 0.00005561 [-0.01538362 to 0.0212081]
  Env-2-ZM96: number analyzed (Participants) | 42 | 42 | 38 | 7
  Env-2-ZM96 | 0.00239069 [-0.0083648 to 0.01101768] | 0.03477023 [0.01804551 to 0.07310345] | 0.034977865 [0.00768028 to 0.11871884] | -0.00905211 [-0.01435048 to 0.00545363]
  LAI Gag: number analyzed (Participants) | 42 | 42 | 38 | 7
  LAI Gag | 0.00479596 [-0.00373824 to 0.01146808] | 0.00389424 [-0.00241976 to 0.01205637] | 0.0069258 [-0.00376213 to 0.0148364] | 0.00050871 [-0.01603156 to 0.0050394]
  LAI gp41TM: number analyzed (Participants) | 42 | 42 | 38 | 7
  LAI gp41TM | -0.006455715 [-0.01597738 to 0.00338559] | -0.00486893 [-0.01386022 to -0.00082034] | -0.00631803 [-0.01802868 to 0.00093287] | -0.00614691 [-0.0264412 to 0.0013653]
  TV1 gp120: number analyzed (Participants) | 42 | 42 | 38 | 7
  TV1 gp120 | 0.064060235 [0.02449973 to 0.16682458] | 0.217194305 [0.13906679 to 0.29238706] | 0.333606595 [0.20594237 to 0.51844985] | -0.00195339 [-0.01595152 to -0.00044574]

11. Primary Outcome: Number of Participants With HIV-specific Total IgG Binding Antibody (Vaccine gp120 Panel) Response Magnitude as Assessed by Binding Antibody Multiplex Assay [Time Frame: Measured at Month 12.]
Description: Serum IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:50 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Values outside the linear range of the assay are not meaningful and are truncated: net MFI less than 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500. Samples from post-enrollment visits have positive responses if: (1) net MFI >= an antigen-specific response threshold (defined as the maximum of 100 and the 95th percentile of baseline net MFI), and (2) net MFI > 3 times baseline net MFI, and (3) experimental antigen MFI > 3 times baseline MFI.
Time Frame: Measured at Month 12
Population: Overall number of participants analyzed represents the HIV uninfected participants with specimens at Month 12. Number Analyzed shows the number of HIV uninfected participants with available BAMA data after filtering for assay specific quality control criteria at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 47 | 45 | 46 | 10
Participants
  1086C_D7gp120.avi/293F at Month 12: number analyzed (Participants) | 47 | 43 | 42 | 9
  1086C_D7gp120.avi/293F at Month 12 | 46 | 43 | 42 | 0
  96ZM651.D11gp120.avi at Month 12: number analyzed (Participants) | 45 | 43 | 43 | 10
  96ZM651.D11gp120.avi at Month 12 | 14 | 22 | 20 | 0
  TV1c8_D11gp120.avi/293F at Month 12: number analyzed (Participants) | 47 | 43 | 43 | 9
  TV1c8_D11gp120.avi/293F at Month 12 | 38 | 43 | 40 | 0

12. Primary Outcome: Level of the HIV-specific Total IgG Binding Antibody (Vaccine gp120 Panel) Response Magnitude as Assessed by Binding Antibody Multiplex Assay [Time Frame: Measured at Month 12.]
Description: Serum IgG responses were measured on a Bio-Plex instrument using a standardized custom Luminex assay, run at 1:50 dilution. The readout is background-subtracted mean fluorescent intensity (MFI), with background adjustment for an antigen-specific plate level control. For each sample, response magnitude is net MFI, defined as experimental antigen MFI minus reference antigen MFI. Values outside the linear range of the assay are not meaningful and are truncated: net MFI less than 1 is set to 1, and net MFI > 22,000 is set to 22,000. Data are excluded if blood draw date was outside the allowable window, a participant was HIV-infected, reference antigen > 5,000 MFI, or baseline net MFI > 6,500.
Time Frame: Measured at Month 12
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 47 | 45 | 46 | 10
relative fluorescence units
  1086C_D7gp120.avi/293F at Month 12: number analyzed (Participants) | 47 | 43 | 42 | 9
  1086C_D7gp120.avi/293F at Month 12 | 7686.25 [3514.25 to 18708.125] | 19787.75 [14907.5 to 22000] | 22000 [22000 to 22000] | 1 [1 to 5]
  96ZM651.D11gp120.avi at Month 12: number analyzed (Participants) | 45 | 43 | 43 | 10
  96ZM651.D11gp120.avi at Month 12 | 938 [491.5 to 2366.75] | 2202.5 [1321.375 to 4108.375] | 2580.5 [1294.375 to 4934.875] | 7.875 [4.0625 to 43.1875]
  TV1c8_D11gp120.avi/293F at Month 12: number analyzed (Participants) | 47 | 43 | 43 | 9
  TV1c8_D11gp120.avi/293F at Month 12 | 1342.75 [658.125 to 5138.875] | 6409.5 [3978.625 to 12420.625] | 8421 [2659.5 to 18775.625] | 1 [1 to 19.75]

13. Secondary Outcome: Occurrence of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine, After the Primary Vaccine Regimen. Measured by Flow Cytometry.
Description: as for outcome 9
Time Frame: Measured at Month 12
Population: In this report, the "overall number of participants analyzed" represents the HIV uninfected participants with specimens at Month12. The "Number Analyzed" in the Outcome Measure Data Table shows the number of participants with available ICS data after filtering for assay specific quality control criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 47 | 45 | 46 | 10
Participants
  1086 gp120: number analyzed (Participants) | 44 | 39 | 40 | 10
  1086 gp120 | 17 | 34 | 33 | 0
  Env-1-ZM96: number analyzed (Participants) | 44 | 39 | 40 | 10
  Env-1-ZM96 | 24 | 34 | 33 | 1
  Env-2-ZM96: number analyzed (Participants) | 44 | 39 | 40 | 10
  Env-2-ZM96 | 2 | 8 | 10 | 0
  LAI Gag: number analyzed (Participants) | 44 | 39 | 40 | 10
  LAI Gag | 0 | 2 | 0 | 0
  TV1 gp120: number analyzed (Participants) | 44 | 39 | 40 | 10
  TV1 gp120 | 24 | 32 | 32 | 0

14. Secondary Outcome: Level of CD4+ T Cell Responses to the HIV Proteins Included in the Vaccine, After the Primary Vaccine Regimen. Measured by Flow Cytometry.
Description: as for outcome 10
Time Frame: Measured at Month 12
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: % CD4+ T-cells
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 47 | 45 | 46 | 10
% CD4+ T-cells
  1086 gp120: number analyzed (Participants) | 44 | 39 | 40 | 10
  1086 gp120 | 0.044319625 [0.009665425 to 0.09187594] | 0.10802498 [0.07815074 to 0.18406719] | 0.15160478 [0.09475396 to 0.30774528] | 0.000078395 [-0.00629445 to 0.00168892]
  Env-1-ZM96: number analyzed (Participants) | 44 | 39 | 40 | 10
  Env-1-ZM96 | 0.060435485 [0.01622735 to 0.085696555] | 0.09662109 [0.05888084 to 0.17217561] | 0.1209486 [0.066832855 to 0.24448282] | 0.00009746 [-0.0063057 to 0.01311592]
  Env-2-ZM96: number analyzed (Participants) | 44 | 39 | 40 | 10
  Env-2-ZM96 | 0.004117915 [-0.002599175 to 0.01463184] | 0.01003653 [0.00256448 to 0.03750046] | 0.020232585 [0.002113855 to 0.040018475] | -0.004564435 [-0.01614768 to -0.00172824]
  LAI Gag: number analyzed (Participants) | 44 | 39 | 40 | 10
  LAI Gag | 0.003934455 [-0.00521375 to 0.007967745] | 0.00199785 [-0.0062505 to 0.00771792] | 0.002998855 [-0.00754884 to 0.01064116] | 0.000049675 [-0.01131992 to 0.00378357]
  TV1 gp120: number analyzed (Participants) | 44 | 39 | 40 | 10
  TV1 gp120 | 0.04961613 [0.01083952 to 0.110185075] | 0.10101452 [0.06202808 to 0.14821607] | 0.145474815 [0.064903025 to 0.24267272] | -0.005495385 [-0.01339975 to -0.00049045]

15. Secondary Outcome: Number of Participants With HIV-specific Total IgG Binding Antibody (Vaccine gp120 Panel) Response Magnitude as Assessed by Binding Antibody Multiplex Assay [Time Frame: Measured at Month 6.5.]
Description: as for outcome 11
Time Frame: Measured at Month 6.5
Population: Overall number of participants analyzed represents the HIV uninfected participants with specimens at Month 6.5. Number Analyzed shows the number of HIV uninfected participants with available BAMA data after filtering for assay specific quality control criteria at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 49 | 48 | 47 | 8
Participants
  1086C_D7gp120.avi/293F at Month 6.5: number analyzed (Participants) | 49 | 45 | 41 | 7
  1086C_D7gp120.avi/293F at Month 6.5 | 49 | 45 | 41 | 0
  96ZM651.D11gp120.avi at Month 6.5: number analyzed (Participants) | 47 | 46 | 41 | 8
  96ZM651.D11gp120.avi at Month 6.5 | 47 | 45 | 39 | 0
  TV1c8_D11gp120.avi/293F at Month 6.5: number analyzed (Participants) | 49 | 46 | 42 | 7
  TV1c8_D11gp120.avi/293F at Month 6.5 | 49 | 46 | 42 | 0

16. Secondary Outcome: Level of the HIV-specific Total IgG Binding Antibody (Vaccine gp120 Panel) Response Magnitude as Assessed by Binding Antibody Multiplex Assay [Time Frame: Measured at Month 6.5]
Description: as for outcome 12
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 49 | 48 | 47 | 8
relative fluorescence units
  1086C_D7gp120.avi/293F at Month 6.5: number analyzed (Participants) | 49 | 45 | 41 | 7
  1086C_D7gp120.avi/293F at Month 6.5 | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 1 [1 to 1]
  96ZM651.D11gp120.avi at Month 6.5: number analyzed (Participants) | 47 | 46 | 41 | 8
  96ZM651.D11gp120.avi at Month 6.5 | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 14.125 [6.375 to 118.8125]
  TV1c8_D11gp120.avi/293F at Month 6.5: number analyzed (Participants) | 49 | 46 | 42 | 7
  TV1c8_D11gp120.avi/293F at Month 6.5 | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 22000 [22000 to 22000] | 1 [1 to 107.625]

17. Secondary Outcome: Area Under Titration Curve of the HIV-specific Total IgG Binding Antibody (Vaccine gp120 Panel) Response Breadth as Assessed by Binding Antibody Multiplex Assay [Time Frame: Measured at Month 6.5.]
Description: Area under titration curve from serial dilution (AUTC) is calculated using the trapezoidal rule based on the raw MFI values truncated at zero across the log base 10 dilution factors, i.e., the summation of products of raw MFI values and log10(dilution factor). The dilution factor refers to the ratio of the volume of the initial (concentrated) solution (V1) to the volume of the final (dilute) solution (V2), and therefore it is unitless. For example, for a dilution of V1:V2=1:50 of a solution, the corresponding dilution factor is V2/V1=50/1=50.
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: RFU*log10(dilution factor)
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 49 | 48 | 47 | 8
RFU*log10(dilution factor)
  1086C_D7gp120.avi/293F at Month 6.5: number analyzed (Participants) | 49 | 45 | 41 | 7
  1086C_D7gp120.avi/293F at Month 6.5 | 40433.144898 [35303.066969 to 44156.283884] | 42528.614697 [41103.049524 to 46165.358075] | 43564.082625 [40648.306087 to 45130.341692] | 0 [0 to 0.1505149978]
  96ZM651.D11gp120.avi at Month 6.5: number analyzed (Participants) | 47 | 46 | 41 | 8
  96ZM651.D11gp120.avi at Month 6.5 | 19137.530429 [12994.975739 to 24038.844376] | 26284.001341 [18696.286306 to 32366.350032] | 19206.42867 [12004.060251 to 26698.726603] | 6.5850311551 [1.2605631068 to 42.962624694]
  TV1c8_D11gp120.avi/293F at Month 6.5: number analyzed (Participants) | 49 | 46 | 42 | 7
  TV1c8_D11gp120.avi/293F at Month 6.5 | 29381.844583 [22547.410076 to 33602.924811] | 36046.799202 [29934.75202 to 39085.348942] | 33717.692497 [26403.115147 to 37738.032754] | 0.0752574989 [0 to 32.30428141]

18. Secondary Outcome: Number of Participants With Anti -V1/V2 Scaffold IgG Binding Antibody ( Vaccine V1V2 Panel) Responses. Measured by Binding Antibody Multiplex Assay (BAMA). [Time Frame: Measured at Month 6.5.]
Description: as for outcome 11
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 49 | 48 | 47 | 8
Participants
  C.1086C_V1_V2 Tags at Month 6.5: number analyzed (Participants) | 48 | 45 | 40 | 8
  C.1086C_V1_V2 Tags at Month 6.5 | 20 | 27 | 19 | 0
  gp70-96ZM651.02 V1v2 at Month 6.5: number analyzed (Participants) | 47 | 45 | 40 | 8
  gp70-96ZM651.02 V1v2 at Month 6.5 | 17 | 24 | 17 | 0
  gp70-TV1.21 V1V2 at Month 6.5: number analyzed (Participants) | 48 | 45 | 40 | 8
  gp70-TV1.21 V1V2 at Month 6.5 | 24 | 26 | 11 | 0
  gp70-TV1.GSKvacV1V2/293F at Month 6.5: number analyzed (Participants) | 47 | 45 | 40 | 8
  gp70-TV1.GSKvacV1V2/293F at Month 6.5 | 29 | 31 | 16 | 0

19. Secondary Outcome: Level of Anti -V1/V2 Scaffold IgG Binding Antibody ( Vaccine V1V2 Panel) Responses. Measured by Binding Antibody Multiplex Assay (BAMA). [Time Frame: Measured at Month 6.5.]
Description: as for outcome 12
Time Frame: Measured at Month 6.5
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 49 | 48 | 47 | 8
relative fluorescence units
  C.1086C_V1_V2 Tags at Month 6.5: number analyzed (Participants) | 48 | 45 | 40 | 8
  C.1086C_V1_V2 Tags at Month 6.5 | 1193.125 [258.5625 to 5013.0625] | 4296.5 [953.25 to 11383] | 1555.5 [381.4375 to 7860.875] | 66.375 [5.5 to 266.9375]
  gp70-96ZM651.02 V1v2 at Month 6.5: number analyzed (Participants) | 47 | 45 | 40 | 8
  gp70-96ZM651.02 V1v2 at Month 6.5 | 429.5 [13 to 2044.875] | 1327.75 [275.25 to 8008.5] | 455.375 [1 to 1275.5625] | 1 [1 to 30]
  gp70-TV1.21 V1V2 at Month 6.5: number analyzed (Participants) | 48 | 45 | 40 | 8
  gp70-TV1.21 V1V2 at Month 6.5 | 209.125 [1 to 1897.0625] | 442.25 [27.75 to 2621.5] | 1 [1 to 543.25] | 1 [1 to 1]
  gp70-TV1.GSKvacV1V2/293F at Month 6.5: number analyzed (Participants) | 47 | 45 | 40 | 8
  gp70-TV1.GSKvacV1V2/293F at Month 6.5 | 225 [1 to 1940.75] | 709.75 [115.75 to 4134.25] | 80.875 [1 to 444.1875] | 1 [1 to 1]

20. Secondary Outcome: Number of Participants With Anti -V1/V2 Scaffold IgG Binding Antibody ( Vaccine V1V2 Panel) Responses. Measured by Binding Antibody Multiplex Assay (BAMA). [Time Frame: Measured at Month 10.]
Description: as for outcome 11
Time Frame: Measured at Month Month 12
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 47 | 45 | 46 | 10
Participants
  C.1086C_V1_V2 Tags at Month 12: number analyzed (Participants) | 47 | 44 | 41 | 10
  C.1086C_V1_V2 Tags at Month 12 | 2 | 3 | 4 | 0
  gp70-96ZM651.02 V1v2 at Month 12: number analyzed (Participants) | 46 | 44 | 42 | 10
  gp70-96ZM651.02 V1v2 at Month 12 | 3 | 4 | 1 | 0
  gp70-TV1.21 V1V2 at Month 12: number analyzed (Participants) | 47 | 44 | 42 | 10
  gp70-TV1.21 V1V2 at Month 12 | 5 | 0 | 2 | 0
  gp70-TV1.GSKvacV1V2/293F at Month 12: number analyzed (Participants) | 46 | 44 | 42 | 10
  gp70-TV1.GSKvacV1V2/293F at Month 12 | 7 | 1 | 2 | 0

21. Secondary Outcome: Level of Anti -V1/V2 Scaffold IgG Binding Antibody ( Vaccine V1V2 Panel) Responses. Measured by Binding Antibody Multiplex Assay (BAMA). [Time Frame: Measured at Month 12.]
Description: as for outcome 12
Time Frame: Measured at Month 12
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: relative fluorescence units
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
Number analyzed (Participants) | 47 | 45 | 46 | 10
relative fluorescence units
  C.1086C_V1_V2 Tags at Month 12: number analyzed (Participants) | 47 | 44 | 41 | 10
  C.1086C_V1_V2 Tags at Month 12 | 90 [23.375 to 264.625] | 235.875 [55.1875 to 502.5] | 153 [60.25 to 471.5] | 18.375 [1.1875 to 99.6875]
  gp70-96ZM651.02 V1v2 at Month 12: number analyzed (Participants) | 46 | 44 | 42 | 10
  gp70-96ZM651.02 V1v2 at Month 12 | 1 [1 to 84.6875] | 1.75 [1 to 258.0625] | 1 [1 to 119.1875] | 1 [1 to 11.1875]
  gp70-TV1.21 V1V2 at Month 12: number analyzed (Participants) | 47 | 44 | 42 | 10
  gp70-TV1.21 V1V2 at Month 12 | 1 [1 to 82.75] | 1 [1 to 30.5] | 1 [1 to 1] | 1 [1 to 1]
  gp70-TV1.GSKvacV1V2/293F at Month 12: number analyzed (Participants) | 46 | 44 | 42 | 10
  gp70-TV1.GSKvacV1V2/293F at Month 12 | 1 [1 to 90.5625] | 1 [1 to 60.8125] | 1 [1 to 11.5] | 1 [1 to 1]

ADVERSE EVENTS:
Time Frame: Serious adverse events are collected throughout the study (months 0-18). Non-serious adverse events are collected through 30 days after each vaccination (at months 0, 1, 3, 6).
Description: Adverse events of special interest (AESI) are defined in Protocol Version 3, Section 6.4.3.2 and Appendix H.
Arm/Group | Vaccine w/ MF59 | Vaccine w/ AS01B - High Dose | Vaccine w/ AS01B - Low Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/10
Other Adverse Events (participants affected / at risk) | 32/50 | 28/50 | 26/50 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine w/ MF59 (N=50) | Vaccine w/ AS01B - High Dose (N=50) | Vaccine w/ AS01B - Low Dose (N=50) | Placebo (N=10)
Any Event in SOC (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Gastrointestinal disorders) | 4 (4) | 1 (1) | 4 (6) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Any Event in SOC (General disorders) | 4 (4) | 5 (7) | 3 (3) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site hypoaesthesia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Infections and infestations) | 19 (23) | 13 (18) | 16 (20) | 2 (3)
Bacterial vaginosis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 6 (8) | 9 (10) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 2 (3) | 2 (2) | 1 (2) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginitis trichomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 4 (5) | 3 (4) | 3 (3) | 0 (0)
Hypobarism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Any Event in SOC (Investigations) | 11 (20) | 13 (26) | 6 (17) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 7 (8) | 4 (5) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (6) | 2 (5) | 3 (8) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 2 (4) | 3 (5) | 0 (0)
Any Event in SOC (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Nervous system disorders) | 4 (4) | 2 (3) | 1 (1) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 5 (6) | 3 (3) | 2 (3) | 1 (1)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 4 (4) | 2 (2) | 2 (3) | 1 (1)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3) | 1 (1) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT03122223/Prot_002.pdf
  • Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT03122223/SAP_003.pdf
  • Informed Consent Form (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT03122223/ICF_000.pdf